CLINICAL TRIAL: NCT02272205
Title: Evaluation of the Effect of a Conventional Antibiotic Prophylaxis on the Positivity of Intraoperative Bacteriological Samples During a Change of Hip or Knee Infected at a Time
Brief Title: Evaluation of Conventional Antibiotic Prophylaxis During a Change of Hip or Knee Infected at a Time
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 004-14
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Total Hip Replacement
Keywords: Hip replacement; Knee replacement; Knee infection; Hip infection; Antibiotic prophylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Retrospective analysis of records

SUMMARY:
Infection is a serious complications after undergoing total hip replacement. It occurs in about 1% of cases. The optimal treatment of these infections is discussed. The team validated by international publications change strategy of the infected prosthesis at a time.

Antibiotic prophylaxis has significantly reduced the infection intraoperative contamination in orthopedic surgery rates. It must be conventionally administered before the surgical incision. In response to infection, it is typically recommended to start this antibiotic after the completion of the deep bacteriological samples, so as not to negate the risk of these samples by the prior administration of antibiotics. This attitude, however, is not formally validated by the scientific literature. In contrast, two recent publications challenge this practice, and suggest the use of a conventional antibiotic prophylaxis even in septic interventions. Our multidisciplinary team opted for a few months for this new strategy. We wish to evaluate the influence of this new approach results in the treatment of infection in total hip or knee.

ELIGIBILITY:
Inclusion Criteria:

* patients operated in service between January 2012 and July 2013 for treatment of an infection of total hip or knee.

Exclusion Criteria:

* patients operated in service before January 2012 and after July 2013 for treatment of an infection of total hip or knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients operated in service between January 2012 and July 2013 for treatment of an infection of total hip or knee.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
concordance of pre-and intraoperative bacteriological documentation | preoperative; intraoperative
  concordance of pre-and intraoperative bacteriological documentation (division into 3 classes: complete, partial, no - Chi-square test

SECONDARY OUTCOMES:
rates to relapse of the initial infection or a new infection | preoperative; intraoperative
  rates to relapse of the initial infection or a new infection (survival curves according to Kaplan-Meier with log-rank test)